CLINICAL TRIAL: NCT04234490
Title: Longitudinal Evaluation of Patient Outcomes and Impact Assessment on Family Members of Home Parenteral Nutrition: New Directions for Research
Brief Title: Longitudinal Evaluation of the Impact of Parenteral Nutrition
Status: Completed | Type: Observational
Sponsor: University of Manchester (Other)
Collaborators: Shire International GmbH (Unknown)
Responsible Party: Principal Investigator, Debra Jones, Nutrition Research Associate, University of Manchester
Other Study IDs: Longitudinal PNIQ
Record Dates: First submitted 2020-01-13; First posted 2020-01-21 (Actual); Last update posted 2022-05-24 (Actual); Status verified 2022-05

CONDITIONS: Parenteral Nutrition
Keywords: Intestinal failure; Quality of life; Carer burden
MeSH Terms: conditions — Hyperphagia; Intestinal Failure | interventions — Parenteral Nutrition; Parenteral Nutrition, Home

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patient: Patients who are receiving Home Parenteral Support (HPN) (artificially fed through a vein) due to intestinal failure
  Interventions: Procedure: Parenteral nutrition
- Carer: Family member or carer of patient who is receiving Home Parenteral Support

INTERVENTIONS:
Procedure: Parenteral nutrition — Impact of parenteral nutrition on patient quality of life over time and impact on carer burden
  Other Names: Home parenteral nutrition, artificial tube feeding
  Groups: Patient

SUMMARY:
Patients with type 3 intestinal failure are completely reliant on artificial feeding and often manage this at home; home parenteral nutrition (HPN). HPN therapy is life saving for these patients.

The Parenteral Nutrition Impact Questionnaire (PNIQ) is a proven tool for measuring quality of life when receiving HPN.

This study will recruit HPN patients across the United Kingdom (UK) and ask them to complete the PNIQ survey at several different time points. This will assess the impact of HPN over time. Family members involved in the participants HPN care will also be asked to complete a carer burden survey (at one time point) to assess the impact of HPN on carers.

DETAILED DESCRIPTION:
Providing a person with food through a vein is known as parenteral nutrition (PN) or artificial tube feeding. This process is used when nutrients from food can't be taken in by the intestine (intestinal failure). Patients with type 3 intestinal failure are completely reliant on artificial feeding and often manage this at home; home parenteral nutrition (HPN). HPN therapy is life saving for these patients.

It is important to assess patients quality of life and their own reported effects of the HPN. The Parenteral Nutrition Impact Questionnaire (PNIQ) is a proven tool for measuring quality of life when receiving HPN.

A recent study involving the use of the PNIQ in multiple hospitals in the UK, showed that those on fewer nights of HPN had better quality of life than those on more nights of HPN. Whilst this was useful for looking at quality of life at one time point, it is now important to assess change in quality life over time and any impact on family members quality of life.

This study will recruit HPN patients across the UK and ask them to complete the PNIQ survey at several different time points. This will assess the impact of HPN over time. Family members involved in the participants HPN care will also be asked to complete a carer burden survey (at one time point) to assess the impact of HPN on carers.

The study is being funded by Shire Pharmaceuticals Ltd.

ELIGIBILITY:
Inclusion Criteria:

Patients:

* All people in receipt of HPN including new patients
* Those 18 years and over.

Carers:

* A family member or person involved in the healthcare of the participating patient. (We will ask patients to nominate their closest family member who in their opinion is potentially most effected by the parenteral feeding.)
* Those 18 years and over.

Exclusion Criteria:

Patients:

* Cannot give informed consent
* Cannot read or write in English.

Carers:

• Family members not directly involved with caring for participants

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Approximately 1400 eligible participants from at least 15 NHS sites who are receiving HPN will be invited to participate. Close family relatives or friends who are carers for the eligible participants will also be invited to participate.
Sampling Method: Probability Sample
Enrollment: 912 (Actual)
Dates: Start 2020-03-02 (Actual); Primary Completion 2022-03-23 (Actual); Study Completion 2022-03-23 (Actual)

PRIMARY OUTCOMES:
Patient reported outcomes | Baseline, five, 10 and 15 months post entry
  Change in Patient reported outcomes (PNIQ score) in people receiving HPN. Score from 0-20, with 0 being high Quality of life and 20 being low quality of life.

SECONDARY OUTCOMES:
Carer burden | Baseline
  Caregiver burden (carer burden survey) in family members/close friends providing HPN healthcare to a patient receiving HPN. Score from 0-84, with 0 being no symptoms and 84 being very severe symptoms
Length of time receiving HPN | Baseline, five, 10 and 15 months post entry
  Amount of time the patient has been receiving HPN (months/years)
Change in number of weekly HPN infusions | Baseline, five, 10 and 15 months post entry
  How often the patient is connected to an infusion each week (numerical)
Change in number of hours connected to HPN infusions each night | Baseline, five, 10 and 15 months post entry
  How many hours the patient is connected to an infusion each night (hours)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Manchester, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Institute research project page — https://www.research.manchester.ac.uk/portal/en/projects/longitudinal-evaluation-of-patient-outcomes-and-impact-assessment-on-family-members-of-home-parental-nutrition-new-directions-for-research(cc9190a3-8571-4b38-a876-a68f1c1eb231).html

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-12-16): https://cdn.clinicaltrials.gov/large-docs/90/NCT04234490/Prot_SAP_000.pdf